CLINICAL TRIAL: NCT02043470
Title: Changes in Regional Retinal Oxygen Extraction and Function After Radiation Therapy
Brief Title: Retinal Oxygen Function After Radiation Therapy
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: UNC Translational and Clinical Sciences (Tracs) (Unknown)
Responsible Party: Sponsor
Other Study IDs: LCCC 1019
Record Dates: First submitted 2014-01-13; First posted 2014-01-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2017-05

CONDITIONS: A History of Radiation Therapy for a Tumor in the Vicinity of the Retina(s)
Keywords: Sinus/nasal cancer
MeSH Terms: conditions — Fistula; Nose Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators propose using retinal oximetry to assess for abnormalities in regional retinal oxygen consumption in previously- irradiated patients, and relate these abnormalities to changes in regional retinal function (i.e. visual field abnormalities). Since different regions of retina receive different radiation doses, the investigators will assess for a dose response as well.

DETAILED DESCRIPTION:
Radiation therapy (RT) is a common treatment for patients with cancers of the sinonasal area, orbit, skull base, nasopharynx, and brain. Because of the close proximity of these targets to the eyes, the retina is often incidentally and unavoidably irradiated. As a result, some patients develop radiation retinopathy and possibly vision loss. Clinicopathologic studies suggest similar microvascular mechanisms for both radiation- and diabetic retinopathy: small vessel occlusion and ischemia that can lead to neovascularization, increased capillary permeability, and visual loss in the regions of retina perfused by damaged vasculature. UNC has a novel, non-invasive retinal imaging technology called a Retinal Oximeter which measures hemoglobin oxygen saturation of retinal vessels. The difference in oxygen saturation between a retinal arteriole and venule pair reflects the oxygen consumption of the retinal region supplied by that vessel pair.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of radiation therapy (no upper age limit)
2. History of radiation therapy delivered at UNC-CH or Rex Hospital to the vicinity of the retina(s) ≥ 2 months prior to enrollment
3. Estimated average dose to at least one quadrant of one retina ≥ 30 Gy

Exclusion Criteria:

1. History of diabetes, retinal vascular occlusions, glaucoma, retinitis pigmentosa, occipital stroke or any other ophthalmologic or systemic problem that may confound visual field results.
2. Residual tumor within the visual pathway: retina, optic nerves, optic chiasm, optic radiations and brain.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a history of radiation therapy for a tumor in the vicinity of the retina(s) at the Department of Radiation Oncology, UNC-CH.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Abnormalities in regional retinal oxygen extraction after incidental irradiation of the retina. | 2 months
  To identify abnormalities in regional retinal oxygen extraction in patients who have had previous incidental irradiation of the retina.
Prevalence of vision loss in patients with previous incidental irradiation of the retina | 2 months
  To determine the prevalence of regional retinal dysfunction (i.e. vision loss) in patients with previous incidental irradiation of the retina.

SECONDARY OUTCOMES:
Changes in retinal oxygen extraction compared to radiation dose | 2 months
  To correlate changes in retinal oxygen extraction to radiation dose.
Vision loss amount versus radiation dose. | 2 months
  To correlate retinal dysfunction (i.e. vision loss) to radiation dose.
Changes in retinal oxygen extraction as compared to vision loss. | 2 months
  To correlate changes in retinal oxygen extraction to retinal dysfunction (i.e. vision loss).

CONTACTS AND LOCATIONS:
Overall Officials: Bhishamjit Chera, MD, Principal Investigator — Department of Radiation Oncology, University of North Carolina Chapel Hill
Locations (1):
- Department of Radiation Oncology Clinic, Chapel Hill, North Carolina, United States